CLINICAL TRIAL: NCT00669526
Title: Clinical and Cost Effectiveness of Brief CBT for Pediatric Internalizing Disorders
Brief Title: Clinical and Cost Effectiveness of Brief Cognitive-Behavioral Therapy (CBT) for Pediatric Internalizing Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); William T. Grant Foundation (Other)
Responsible Party: V. Robin Weersing, Ph.D. / Principal Investigator, SDSU/UCSD Joint Doctoral Program in Clinical Psychology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 051653
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Depression; Anxiety
Keywords: anxiety; depression; Major Depressive Disorder; child; adolescent; CBT; Cognitive-Behavioral Therapy; primary care
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMHC referral (Active Comparator): Referral to local Specialty Mental Health Care Services
  Interventions: Behavioral: SMHC referral
- BCBT (Experimental): Brief Cognitive Behavioral Therapy
  Interventions: Behavioral: BCBT

INTERVENTIONS:
Behavioral: BCBT — Brief Cognitive Behavioral Therapy. This BCBT protocol consists of up to 8 CBT sessions to be conducted over a maximum of 12 weeks.
  Other Names: CBT; Cognitive-Behavioral Therapy
  Arms: BCBT
Behavioral: SMHC referral — Referral to local Speciality Mental Health Care. Families were referred to local mental health care providers, and could freely choose any treatment or combination of treatments offered (e.g., anti-depressant medication, individual psychotherapy, family psychotherapy, etc.).
  Arms: SMHC referral

SUMMARY:
This project assesses the clinical and cost effectiveness of brief cognitive-behavioral therapy (CBT) for depressed (ages 11-17) and anxious (ages 8-17) youths seen for services in pediatric primary care. This study is designed to compare the impact of brief CBT delivered on-site in pediatric primary care to referral to specialty mental health care (SMHC), as well as obtain an estimate of the total costs of the CBT protocols for depression and anxiety and the cost-effectiveness of the protocols compared to referral to and utilization of SMHC services.

ELIGIBILITY:
Inclusion Criteria for depression:

* Ages 11 to 17 years
* Meet diagnostic criteria for Major Depression, Dysthymia, or Minor Depression
* Live with a legal guardian

Inclusion Criteria for anxiety:

* Ages 7 to 17 years
* Meet full or probable (missing one, non-core symptom) diagnostic criteria for Separation Anxiety Disorder, Generalized Anxiety Disorder, Social Phobia, or Specific Phobia
* Live with a legal guardian

Exclusion Criteria:

* Require treatment other than brief CBT (namely, youths with bipolar disorder, psychosis, active suicidal ideation with plan, post-traumatic stress disorder, substance dependence, or mental retardation
* Experience of recent physical or sexual maltreatment
* Serious or unstable physical illness
* Current participation in an alternate, active intervention for the target condition of interest

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2004-10; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Clinician Global Impressions - Improvement (CGI-I) | weeks 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: V. Robin Weersing, Ph.D., Principal Investigator — SDSU/UCSD Joint Doctoral Program in Clinical Psychology
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Weersing, V. R., Gonzalez, A., Campo, J. V., & Lucas, A. N. Brief Behavioral Therapy for Pediatric Anxiety and Depression: Piloting an Integrated Treatment Approach. Cognitive and Behavioral Practice (in press), 2008.
- See also: The National Institute of Mental Health (NIMH) is the largest scientific organization in the world dedicated to research focused on the understanding, treatment, and prevention of mental disorders and the promotion of mental health. — http://www.nimh.nih.gov/
- See also: The Robert Wood Johnson Foundation (RWJF) focuses on the pressing health and health care issues facing our country. — http://www.rwjf.org/
- See also: William T. Grant Foundation's mission focuses on improving the lives of youth ages 8 to 25 in the United States. We accomplish this by providing grants primarily for high-quality empirical studies. — http://www.wtgrantfoundation.org/